CLINICAL TRIAL: NCT06729710
Title: Prism Adaptation in Symptomatic Esophoria - Effect of Shorter Time Intervals and Surgical Outcomes Based on Prism Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mikael Hofsli, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24017032
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Esophoria
Keywords: Esophoria; prism adaptation; strabismus surgery
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 hour prism adaptation (Active Comparator): Patients who receive one hour of prism adaptation.
  Interventions: Procedure: Prism adaptation test; Procedure: other
- 4 hours of prism adaptation (Active Comparator): Patients who receive four hour of prism adaptation.
  Interventions: Procedure: Prism adaptation test; Procedure: other

INTERVENTIONS:
Procedure: Prism adaptation test — Prism Adapation test for 1 hour in one group, and 4 hours in second group
Procedure: other — Surgery based on prism adaptation test of 1 hour in one group and 4 hours in second group
  Other Names: Surgery based on prism adaptation test

SUMMARY:
This study is a prospective randomized study aiming to investigate the effect of prism adaptation before surgery for symptomatic esophoria on the number of reoperations, the occurrence of over- and under-correction after the first surgery, and symptom resolution. Additionally, we aim to define the optimal duration of prism adaptation.

DETAILED DESCRIPTION:
SUBSTUDY 1 The Optimal Duration of Prism Adaptation in Symptomatic Esophoria Study Design: Prospective, randomized controlled study Patient Group: 100 participants with symptomatic esophoria, randomized into two groups of 50 participants each to undergo either one hour or four hours of prism adaptation.

The purpose of this study is to determine the optimal duration of prism adaptation.

The hypothesis is that the measured deviation angle is expected to increase after one hour of prism adaptation compared to before prism adaptation. Furthermore, it is expected that the measured deviation angle will not differ significantly between the two randomization groups. The primary endpoint is the measured deviation angle at the conclusion of prism adaptation.

The results are highly relevant for accurate surgical dosing (and thus postoperative symptoms and reoperation rates), efficient use of hospital resources, and reduced patient waiting times in the outpatient clinic.

SUBSTUDY 2 Strabismus Surgery for Symptomatic Esophoria Based on Prism Adaptation Study Design: Prospective, randomized controlled study Patient Group: 100 participants with symptomatic esophoria, using the same patients and randomization groups as in Substudy 1.

The purpose of this study is to investigate the effectiveness of strabismus surgery for symptomatic esophoria based on prism adaptation. Patients randomized in Substudy 2 to either one or four hours of prism adaptation will undergo surgery based on the full prism-adapted angle.

The hypothesis for this substudy is that surgical dosing based on one hour of prism adaptation will be equivalent to dosing based on four hours of prism adaptation. The primary endpoint will be the reoperation rate. Secondary endpoints will include comparisons of preoperative surgical planning metrics (target deviation and number of eye muscles operated), symptom resolution after the first surgery, and prism measurements (including rates of over- and undercorrections).

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic esophoria who meet one or more of the following criteria:

* Double vision
* Asthenopia (eye strain)
* Headaches related to esophoria
* Worsening of symptoms during fatigue, sleep deprivation, reading, illness, or alcohol consumption.

Exclusion Criteria:

* Age between 18 and 65 years at date of inclusion.
* Accommodative esotropia or esophoria
* Myopia exceeding 10 diopters in the most myopic meridian
* Treatment with botulinum toxin in an eye muscle within four months prior to inclusion
* Inability to undergo reliable orthoptic measurements or prism adaptation
* Previous strabismus surgery
* Pregnancy or breastfeeding within 12 months prior to inclusion
* Myogenic disorders (including Myasthenia Gravis)
* Restrictive strabismus (including previous eye muscle trauma or Graves' orbitopathy)
* Eye muscle paresis
* Maximum prism-adapted deviation angle >40 prism diopters (PD) in any gaze direction for distance
* Maximum prism-adapted deviation angle with ≥20 PD difference between near and distance measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Reoperation rate | Up to 5 years
  Number of patients in need of reoperation after initial surgery for symptomatic esophoria
Measured deviation angle at the conclusion of prism adaptation. | Up to 5 years
  Measured deviation angle in prism diopters at the conclusion of prism adaptation.

SECONDARY OUTCOMES:
Motor success | 1 year from date of surgery
  Motor success: 10 prism diopters of esophoria to 5 prism diopters of exophoria measured with prism alternating cover test.
  Motor failure: Manifest strabismus measured with prism alternating cover test
Sensory success | 1 year from date of surgery
  Sensory success: Postoperative unchanged or improvement in stereopsis measured in seconds of arc with the same method (LANG I/II or TNO) in compared to baseline.
Symptomatic success | 1 year from date of surgery
  Symptomatic success: Single vision (defined as the absence of double vision in daily life) and/or absence of asthenopia (defined as eye strain that is significant in daily life)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No